CLINICAL TRIAL: NCT06342765
Title: Safety and Performance of the SpineVision Posterior Fixation Systems Lumis®, Plus® and Ulis® in Thoracolumbar Spinal Degenerative Pathologies or Degenerative Disc Disease (DDD) Associated Pathologies Treatment - Fixed D3 Study
Brief Title: Safety and Performance of the SpineVision Posterior Fixation Systems in Thoracolumbar Spinal Treatment
Acronym: FixedD3
Status: Recruiting | Type: Observational
Sponsor: SPINEVISION SAS (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Other Study IDs: SV009
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Intervertebral Disc Degeneration
Keywords: Lumbar; Spine; Fusion; Posterior fixation; Oswestry disability index; Visual Analogue Score
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Pedicle fixation surgery — Pedicle fixation surgery indicates a surgical approach in the thoracic spine down to sacral spine to either support interbody fusion (fusion of the discal space between two vertebrae) , or to correct spinal deformity.

SUMMARY:
The goal of this observational study is to confirm the safety and performance of the three (3) Spinevision posterior fixations systems Lumis®, Plus® and Ulis® , in the treatment of patient suffering from thoracolumbar spinal degenerative pathologies, or degenerative disc disease (disease that occurs when the spinal disk break down) associated pathologies.

Part of their standard of care, participants will be questioned on their back and leg pains, their disability and if they have encountered any adverse effects since the Spinevision posterior fixation system implant surgery. Those data will be collected up to twenty four (24) months after the Spinevision posterior fixation system implant surgery.

DETAILED DESCRIPTION:
The Fixed D3 study is a multicentric, non-randomized, ambispective, post market clinical follow-up study. This means that either subjects already implanted with one (1) of the Spinevision posterior fixations systems (Lumis, Plus or Ulis) - retrospective subjects - or subjects planned for treatment with one of the Spinevision posterior fixation system (prospective subjects) can be enrolled in the study.

Standard of care data up to twenty four (24) months post Spinevision posterior fixation system implant procedure will be collected; key data include back and leg Visual Analogue Score (VAS) pain, Oswestry Disability Index (ODI) score, and adverse events.

Data will be collected at pre-operative, per-operative, and post-operative Month 2, Month 6, Month 12 and Month 24.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with Lumis®, Plus® or Ulis® posterior fixation system
* Patient of 18 years old and more
* Patient has provided signed informed consent or did not oppose to his/her data collection, per local regulation

Exclusion Criteria: contra-indication

* trauma (i.e., fracture or dislocation)
* Known or suspected allergy or intolerance to the implanted material, mainly to metal (e.g., cobalt, chromium, nickel, etc.)
* Any other medical or surgical condition likely to compromise the success of instrumented surgery, such as the presence of a malignant tumor or serious congenital abnormalities, raised erythrocyte sedimentation rate not explained by other diseases, high white blood cell count or a tendency to low white blood cell count
* All cases not described in the indications
* Localized infection of the operative site
* All patients with insufficient tissue cover of the operative site
* Local signs of inflammation
* Fever or leukocytosis
* Pathological obesity
* Pregnancy
* Mental illness
* Rapidly evolving joint diseases, bone absorption, osteopenia and/or osteoporosis. Osteoporosis is a relative contraindication, as this medical condition can limit the expected correction gain and stability of mechanical fixation
* All cases not requiring bone graft or bone fusion
* When pedicular screws are used, absence or malformation of pedicles
* All cases requiring a combination of different metals
* All patients not agreeing to comply with post-operative instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for treatment or already treated with one (1) of the SpineVision posterior fixation system (Lumis®, Plus® or Ulis®) will be offered to participate in the study; this applies to primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious and non-serious device- and/or procedure-related adverse events | Month 24
  Rate of the serious and non-serious device- and/or procedure-related adverse events will be analyzed and compared to the state of the art.
Change of the Oswestry Disability Index (ODI) | Month 12
  Oswestry Disability Index (ODI) mean score at Month 12 will be compared to the ODI mean score at baseline.

SECONDARY OUTCOMES:
Fusion success | Month 2, month 6, month 12 and month 24
  Fusion rate will be analyzed and compared to the state if the art.
Change of the Oswestry Disability Index (ODI) | Month 2, month 6, month 12 and month 24
  Mean Oswestry Disability Index (ODI) score evolution score will be analyzed.
Change of the back and leg Visual Analogue Score (VAS) | Month 2, month 6, month 12 and month 24
  Back and leg Visual Analogue Score (VAS) pain assessment will be analyzed.
Incidence of revision surgery at implant site | Month 2, month 6, month 12 and month 24
  Rate of revision surgery at implant site will be analyzed and compared to the state of the art.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pommier, Principal Investigator — Orthéo Neurochirurgie
Locations (3):
- France (3):
  - DOSCEA Pôle Rachis, Bayonne
  - Clinique du dos Bordeaux-Terrefort, Bruges
  - Orthéo Neurochirurgie, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No